CLINICAL TRIAL: NCT00591812
Title: Evaluation of the Compress Distal Femoral Replacement System
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 00-038
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Lower Thighbone and Knee Joint Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 - ComPreSs system (Experimental)
  Interventions: Device: ComPreSs Distal Femoral Replacement System.

INTERVENTIONS:
Device: ComPreSs Distal Femoral Replacement System. — ComPreSs system of intramedullary fixation along with the Finn Knee system

SUMMARY:
Patients in this study require a replacement of a lower thighbone and knee joint. A new device, called the ComPreSs, will be used in this study to replace the lower thighbone. This new device has not yet been approved by the Food and Drug Administration (FDA). There is not enough data to assure that it is as good as other devices currently available. Taking part in this study will help provide data to the FDA. Other devices used to replace large pieces of bone and joints in the leg can result in damage to the bone over time. The bone damage can cause the device to come loose from the bone. This is a bad problem, and causes pain, and often more surgery is needed. This new device connects to the bone in a different way to prevent some of the problems seen with other devices. The new device protects the bone, and may help the replacement last longer. So far, the device has been used in over 50 patients on a selective basis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bone tumors of the distal femur requiring primary bone resection of up to 30 cm with the resection at or below the lesser trochanter.
* Patients with prior orthopaedic oncologic conditions requiring revisions of distal femoral replacement devices with a total replacement height of 30 cm or less and the resection level is at or below the lesser trochanter.
* Patients who have a cortical bone thickness of 2.5 mm or larger in the region where the ComPreSs device would be implanted.
* Patients diagnosed with a bone tumor classified as Stage 1A, IB, IIA, IIB, or III by Enneking's classification system. (See section 12.0, #7)

Exclusion Criteria:

* Patients with active infection.
* Patients who are unable to return for follow-up examinations.
* Patients who have cortical bone thickness less than 2.5 mm in the region where the ComPreSs device would be implanted.
* Patients who are unwilling or incapable of following postoperative care instructions.
* Patients requiring bilateral knee implants.
* Patients with evidence of vascular insufficiency (arterial and/or venous).
* Patients having Parkinson's disease, severe muscular atrophy, neuromuscular disease in the affected limb.
* Patients with prior irradiated bone.
* Patients with metastatic cancer including carcinoma, melanoma, myeloma, lymphoma, leukemia.
* Patients with pathologic soft tissue or skeletal conditions that would prevent secure fixation of the device in the bone.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2000-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Healey, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/